CLINICAL TRIAL: NCT05535959
Title: A Phase 1, Randomized, Open-label, Crossover Study to Evaluate the Relative Bioavailability of a Fixed-dose Combination Tablet of VX-121, Tezacaftor, and Deutivacaftor in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Relative Bioavailability of a Fixed-dose Combination Tablet of VX-121/Tezacaftor/Deutivacaftor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VX22-121-009
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Participants will receive a single dose of reference FDC tablet of VX-121/TEZ/D-IVA in dosing period 1, followed by a single dose of test FDC tablet of VX-121/TEZ/D-IVA in dosing period 2. A washout period of 14 days will be maintained between the 2 dosing periods.
  Interventions: Drug: VX-121/TEZ/D-IVA
- Sequence 2 (Experimental): Participants will receive a single dose of test FDC tablet of VX-121/TEZ/D-IVA in dosing period 1, followed by a single dose of reference FDC tablet of VX-121/TEZ/D-IVA in dosing period 2. A washout period of 14 days will be maintained between the 2 dosing periods.
  Interventions: Drug: VX-121/TEZ/D-IVA

INTERVENTIONS:
Drug: VX-121/TEZ/D-IVA — FDC tablet for oral administration.
  Other Names: VX-121/VX-661/CTP-656; VX-121/VX-661/VX-561; VX-121/tezacaftor/deutivacaftor

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of a fixed-dose combination tablet (FDC) of VX-121/tezacaftor/deutivacaftor (VX-121/TEZ/D-IVA).

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (Kg/m^2), both inclusive
* A total body weight greater than (>)50 kg

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption
* Female participants who are pregnant, nursing, or planning to become pregnant during the study or 90 days after the last dose of the study drug
* Male participants with a female partner who is pregnant, nursing, or planning to become pregnant during the study
* History of cardiovascular disease or central nervous system disease

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of VX-121, TEZ, and D-IVA | Pre-dose up to 288 hours Post-dose
Area Under the Concentration Versus Time Curve (AUC) of VX-121, TEZ, and D-IVA | Pre-dose up to 288 hours Post-dose

SECONDARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Salt Lake City, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing